CLINICAL TRIAL: NCT03202329
Title: Evaluation of Post-operative, Nurse-based Heart Failure Care Compared to Standard Treatment in Patients With Heart Failure Undergoing Non-cardiac Surgery
Brief Title: Evaluation of Post-operative, Nurse-based Heart Failure Care in Non-cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Birgit Assmus (Other)
Responsible Party: Sponsor-Investigator, Birgit Assmus, Prof. Dr. med., Johann Wolfgang Goethe University Hospital
Organization: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HFS-01
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure，Congestive
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Other): responsible surgeon has actively to ask for cardiology support (he decides whether a heart failure specialist should see the patient post-operatively)
  Interventions: Other: standard care
- nurse-based care (Other): heart failure nurses visit postoperatively every (working-) day to check fluid balance, medication, rhythm and general condition
  Interventions: Other: Nurse-based care

INTERVENTIONS:
Other: standard care — cardiologists assist in treatment and provide heart failure guidance post-operatively if required by the treating surgeon
  Arms: standard care
Other: Nurse-based care — board-certified heart failure nurses provide heart failure guidance post-operatively on every working day
  Arms: nurse-based care

SUMMARY:
Patients with heart failure NYHA >= II receiving non-emergent non-cardiac in-patient surgery will be randomized to receive either standard post-operative care (surgeon has to ask actively for specialist cardiological support) or a nurse-based heart failure management (nurses provide week-day support every day after surgery, if needed together with a heart failure doctor)

ELIGIBILITY:
Inclusion Criteria:

patients with heart failure NYHA >= II (HFrEF and HFpEF) or LVEF <= 40% non-cardiac surgery planned later than 24 hours age > 18 years written informed consent

Exclusion Criteria:

patients on intensive care life-expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
composite endpoint of in-hospital heart failure-related complications (readmission on ICU, re-initiation of inotropic support, pleural effusion, pulmonary edema, pneumonia requiring antibiotic treatment, non-invasive or invasive ventilation) | 30 days
  severe heart-failure related clinical events during hospitalisation for non-cardiac surgery

SECONDARY OUTCOMES:
days in hospital | 90 days
  total days in hospital for non-cardiac surgery
acute kidney injury | 90 days
  Acute kidney injury grade: 0 = Creatinine increase < 1,5 x baseline, Stage 1 Creatinine increase > 1,5 x baseline, Stage 2 Creatinine increase > 2 x baseline, Stage 3 Creatinine increase > 3 x baseline)
Qulity of Life by SF-12 | 90 days
  repetitive assessment with SF-12

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Goethe University Hospital, Frankfurt am Main, Hesse
  - Klinikum Goethe University, Frankfurt am Main

IPD SHARING:
Plan to Share IPD: Undecided